CLINICAL TRIAL: NCT06581497
Title: Comparing the Efficacy of ICIs With and Without MWA in Advanced Hepatocellular Carcinoma in Real-World Clinical Practice
Brief Title: ICIs With and Without MWA in Advanced Hepatocellular Carcinoma
Acronym: IMI-aHCC
Status: Completed | Type: Observational
Sponsor: The First People's Hospital of Neijiang (Other)
Responsible Party: Principal Investigator, Ou Jiang, Director of Cancer Center, Neijiang No.2 People's Hospital
Other Study IDs: 2026RP-0106-03
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: HCC; Therapy Adverse Effect
Keywords: HCC; anti-PD-1 mAbs; thermal ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICIs: ICIs mainly refer to PD-1 drug therapy, including pembrolizumab, camrizumab, toripalimab, tislelizumab, and sintilimab. The dosage and duration of ICIs comply with the manufacturer's guidelines.
  Interventions: Drug: ICIs
- MWA+ICIs: ICIs mainly refer to PD-1 drug therapy, including pembrolizumab, camrizumab, toripalimab, tislelizumab, and sintilimab. The dosage and duration of ICIs comply with the manufacturer's guidelines. All patients, except for those enrolled in ICIs, should also undergo MWA treatment.
  Interventions: Procedure: ICIs+MWA

INTERVENTIONS:
Drug: ICIs — ICIs mainly refer to PD-1 drug therapy, including pembrolizumab, camrizumab, toripalimab, tislelizumab, and sintilimab. The dosage and duration of ICIs comply with the manufacturer's guidelines.
  Groups: ICIs
Procedure: ICIs+MWA — ICIs mainly refer to PD-1 drug therapy, including pembrolizumab, camrizumab, toripalimab, tislelizumab, and sintilimab. The dosage and duration of ICIs comply with the manufacturer's guidelines. All patients, except for those enrolled in ICIs, should also undergo MWA treatment.
  Groups: MWA+ICIs

SUMMARY:
Immunotherapy has become the main treatment recommendation for HCC. MWA treatment induces peripheral immune response, which may enhance the effectiveness of immunotherapy for advanced HCC. This study aims to compare the efficacy and safety of ICIs combined with MWA compared to ICIs alone.

The study will compare two groups: ICIs and ICIs+MWA. Main objectives: OS, PFS Secondary objectives: CR PR、SD、PD、ORR、DCR、AEs This study addresses the efficacy and safety of using ICIs in combination with MWA compared to ICIs alone for advanced HCC patients.

The investigators' study aims to evaluate the necessity of immunotherapy combined with targeted drugs or microwave ablation in patients with advanced hepatocellular carcinoma in the real world, providing relevant clinical data for the treatment selection of HCC patients.

DETAILED DESCRIPTION:
Research Title: Comparing the Efficacy of ICIs with and without MWA in Advanced Hepatocellular Carcinoma in Real Clinical Practice Background: Immunotherapy has become the main treatment recommendation for cancer. Ablation therapy induces peripheral immune response, which may enhance the effectiveness of immunotherapy in patients with advanced hepatocellular carcinoma (HCC).

Main objectives: OS, PFS Secondary objectives: CR PR、SD、PD、ORR、DCR、AEs Research Design: This is a single center, retrospective cohort study. This study addresses the efficacy and safety of using ICIs in combination with MWA compared to ICIs alone for advanced HCC patients.

Meaning: The investigators' study aims to evaluate the necessity of immunotherapy combined with targeted drugs or microwave ablation in patients with advanced hepatocellular carcinoma in the real world, providing relevant clinical data for the treatment selection of HCC patients.

Innovation: The innovation of this paper lies in the first verification of the efficacy and safety of microwave ablation (MWA) combined with immune checkpoint inhibitors (ICIs) in the treatment of advanced hepatocellular carcinoma (HCC) patients.

Expected results: The innovation of this paper lies in the first validation of the significant efficacy of microwave ablation (MWA) combined with immune checkpoint inhibitors (ICIs) in the treatment of advanced hepatocellular carcinoma (HCC) patients, significantly improving overall survival (OS) and progression free survival (PFS), as well as objective response rate (ORR) and disease control rate (DCR).

Conclusion: The investigators' study aims to evaluate the necessity of immunotherapy combined with targeted drugs or microwave ablation in patients with advanced hepatocellular carcinoma in the real world, providing relevant clinical data for the treatment selection of HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Gender is not limited, age range is 19-80 years old.
* Meets the clinical diagnostic criteria for HCC.
* Progress after first-line treatment.
* CNLC staging: Stage IIa, IIb, or IIIb of advanced HCC.
* Child Pugh liver function grading score 5-7 points.
* The ECOG (Eastern Cooperative Oncology Group) score ranges from 0 to 1.
* The patient has a certain degree of compliance with the treatment plan and follow-up performance.
* For patients infected with hepatitis B, antiviral treatment with anti hepatitis B virus drugs should be carried out before receiving treatment; And the hepatitis B DNA titer of the patient was less than 10^2 IU/ml.

Exclusion Criteria:

* It has been determined that the inclusion criteria cannot be met.
* Enhanced CT or MRI shows more than 3 active lesions in the liver, and the shortest diameter of a single lesion is greater than 3cm.
* There is a portal vein cancer thrombus present.
* The extrahepatic metastatic lesions have not been well controlled.
* Other treatments were received during the process of receiving immunotherapy or immunotherapy combined with MWA treatment.
* There is active bleeding present.
* There are interstitial lung diseases, pulmonary fibrosis, and autoimmune diseases present.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators applied inclusion criteria, requiring a score of 0-1 for the Eastern Cooperative Oncology Group Performance Status (ECOG PS), The study includes patients in BCLC phases B and C, classified as Child Pugh A or B (score ≤ 7 points), with an expected lifespan of at least 3 months. Other inclusion criteria are liver function ≤ twice the upper limit of the normal value, creatinine ≤ 1.5 times the upper limit of the normal value, serum albumin level > 25 g/L, platelet count > 50 × 10^9/mm³, precursor activity > 50%, total white blood cell count > 1.5 × 10^9/mm³, and hemoglobin level > 80 g/m³. Primary exclusion criteria include interstitial lung disease, pulmonary fibrosis, autoimmune disease, and a history of liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Progression-Free Survival was assessed from the date of treatment initiation until the date of first documented disease progression or death from any cause, whichever occurred first, assessed up to 24 months.
  Time from treatment initiation to disease progression or death from any cause.
Overall Survival (OS) | Overall Survival was measured from the date of treatment initiation until death from any cause or patients who were still alive at the last follow-up were censored at that time point, assessed up to 36 months.
  Time from treatment initiation to disease progression or death from any cause.

SECONDARY OUTCOMES:
objective response rate (ORR) | Objective response rate was measured from baseline to 24 months, every 8 weeks or until disease progression, unacceptable toxicity, or withdrawal from the study, whichever occurs first.
  According to the mRECIST criteria, the proportion of patients who achieve complete response (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Neijiang City, Neijiang, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grandhi MS, Kim AK, Ronnekleiv-Kelly SM, Kamel IR, Ghasebeh MA, Pawlik TM. Hepatocellular carcinoma: From diagnosis to treatment. Surg Oncol. 2016 Jun;25(2):74-85. doi: 10.1016/j.suronc.2016.03.002. Epub 2016 Mar 5. PMID 27312032
- [Background] McGuire S. World Cancer Report 2014. Geneva, Switzerland: World Health Organization, International Agency for Research on Cancer, WHO Press, 2015. Adv Nutr. 2016 Mar 15;7(2):418-9. doi: 10.3945/an.116.012211. Print 2016 Mar. No abstract available. PMID 26980827
- [Background] Zhou Y, Xu X, Ding J, Jing X, Wang F, Wang Y, Wang P. Dynamic changes of T-cell subsets and their relation with tumor recurrence after microwave ablation in patients with hepatocellular carcinoma. J Cancer Res Ther. 2018 Jan;14(1):40-45. doi: 10.4103/jcrt.JCRT_775_17. PMID 29516957
- [Background] Zhang H, Hou X, Cai H, Zhuang X. Effects of microwave ablation on T-cell subsets and cytokines of patients with hepatocellular carcinoma. Minim Invasive Ther Allied Technol. 2017 Aug;26(4):207-211. doi: 10.1080/13645706.2017.1286356. Epub 2017 Feb 20. PMID 28635405
- [Background] Khan AA, Liu ZK, Xu X. Recent advances in immunotherapy for hepatocellular carcinoma. Hepatobiliary Pancreat Dis Int. 2021 Dec;20(6):511-520. doi: 10.1016/j.hbpd.2021.06.010. Epub 2021 Jul 24. PMID 34344612
- [Background] Brown ZJ, Greten TF, Heinrich B. Adjuvant Treatment of Hepatocellular Carcinoma: Prospect of Immunotherapy. Hepatology. 2019 Oct;70(4):1437-1442. doi: 10.1002/hep.30633. Epub 2019 Sep 19. PMID 30927283
- [Background] van den Bijgaart RJ, Eikelenboom DC, Hoogenboom M, Futterer JJ, den Brok MH, Adema GJ. Thermal and mechanical high-intensity focused ultrasound: perspectives on tumor ablation, immune effects and combination strategies. Cancer Immunol Immunother. 2017 Feb;66(2):247-258. doi: 10.1007/s00262-016-1891-9. Epub 2016 Sep 1. PMID 27585790
- [Background] Fatourou EM, Koskinas JS. Adaptive immunity in hepatocellular carcinoma: prognostic and therapeutic implications. Expert Rev Anticancer Ther. 2009 Oct;9(10):1499-510. doi: 10.1586/era.09.103. PMID 19828011
- [Background] Rao P, Escudier B, de Baere T. Spontaneous regression of multiple pulmonary metastases after radiofrequency ablation of a single metastasis. Cardiovasc Intervent Radiol. 2011 Apr;34(2):424-30. doi: 10.1007/s00270-010-9896-9. Epub 2010 Jun 8. PMID 20532778
- [Background] Huang ZM, Lai CX, Zuo MX, An C, Wang XC, Huang JH, Ning E. Adjuvant cytokine-induced killer cells with minimally invasive therapies augmented therapeutic efficacy of unresectable hepatocellular carcinoma. J Cancer Res Ther. 2020;16(7):1603-1610. doi: 10.4103/jcrt.JCRT_962_19. PMID 33565506